CLINICAL TRIAL: NCT01919411
Title: Prophylactic Antibiotics After Functional Endoscopic Sinus Surgery: a Randomized, Double-blind Placebo Controlled Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Responsible Party: Principal Investigator, Eric Holbrook, Principal Investigator, Massachusetts Eye and Ear Infirmary
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11-053H
Record Dates: First submitted 2013-08-01; First posted 2013-08-09 (Estimated); Results first posted 2020-02-10 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Sinusitis
Keywords: Chronic rhinosinusitis; Sinus surgery; Antibiotics
MeSH Terms: conditions — Sinusitis | interventions — Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Amoxicillin-Potassium Clavulanate (Experimental): All patients in the study will undergo endoscopic sinus surgery. This arm will receive 7 days of augmentin (amoxicillin-clavulanate) 500mg orally twice a day after surgery.
  Interventions: Drug: Amoxicillin-Potassium Clavulanate
- Placebo (Placebo Comparator): All patients in the study will undergo endoscopic sinus surgery. This arm will receive 7 days of placebo orally twice a day after surgery.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Amoxicillin-Potassium Clavulanate — Patients in this arm will receive 500mg of Amoxicillin-Potassium Clavulanate Combination orally twice a day for 7 days after surgery.
  Other Names: Augmentin
  Arms: Amoxicillin-Potassium Clavulanate
Drug: Placebo — Patients in this arm will receive 7 days of placebo after surgery.
  Arms: Placebo

SUMMARY:
Surgeons commonly prescribe post operative prophylactic antibiotics after sinus surgery. There is minimal data to support this. The investigators' study will aim to demonstrate that patients' quality of life and rate of post operative infection is the same whether they receive or do not receive antibiotics post operatively. The investigators hypothesis is that the disease specific quality of life of patients taking post-operative antibiotics is not inferior to the quality of life of patients who do not take post-operative antibiotics, and the rate of post-operative infections are the same. The investigators' specific aim is to compare validated symptom scores between post-operative populations who are given or are not given antibiotics. Rates of infections in the first 10 days after surgery will be recorded. The investigators will also compare endoscopic grades of sinus cavities during the post-operative follow up exams as an additional outcome measure.

DETAILED DESCRIPTION:
Functional endoscopic sinus surgery (FESS) is a commonly performed procedure in the United States to treat chronic rhinosinusitis. Common practice is to prescribe prophylactic antibiotics postoperatively. This is similar to the long tradition of prophylactic antibiotics after tonsillectomy. The American Academy of Otolaryngology - Head and Neck Surgery recently strongly recommended against prophylactic antibiotics after tonsillectomy. In this light, this study would demonstrate the lack of need for antibiotics after FESS. Currently one surgeon does not prescribe antibiotics except when evidence of active infection was found during surgery. The other surgeon in the study currently prescribes antibiotics. This study would prospectively compare the two groups in a randomized fashion. The investigators' plan to use the Sinonasal outcomes test - 22 (SNOT-22) as the investigators' primary outcomes measure, which is a validated quality of life instrument in sinusitis.

ELIGIBILITY:
Inclusion Criteria:

- Patients eligible for surgery would be patients with chronic rhinosinusitis (defined by the AAOHNS 2007 consensus statement by Rosenfeld et al) and have been determined by their surgeons to have persistent symptoms after maximal medical therapy. Maximal medical therapy is defined as a course of broad spectrum or culture-directed antibiotics used in conjunction with a nasal steroid.

Exclusion Criteria:

1. Penicillin, cephalosporin, amoxicillin/clavulanate allergy
2. Cystic Fibrosis
3. Immunodeficiency
4. Presence of any foreign body (ie.absorbable and non-absorbable packing) after surgery
5. Odontogenic causes of sinusitis
6. Fungal ball
7. Infected mucocele
8. Complication of sinusitis (meningitis, orbital complication, cellulitis, brain abscess)
9. Non endoscopic sinus surgery (Caldwell luc, external approaches, etc)
10. Age <18
11. Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2013-02; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric H Holbrook, MD, Principal Investigator — MEEI
Locations (1):
- Massachusetts Eye and Ear Infirmary, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hopkins C, Gillett S, Slack R, Lund VJ, Browne JP. Psychometric validity of the 22-item Sinonasal Outcome Test. Clin Otolaryngol. 2009 Oct;34(5):447-54. doi: 10.1111/j.1749-4486.2009.01995.x. PMID 19793277
- [Background] Rosenfeld RM, Andes D, Bhattacharyya N, Cheung D, Eisenberg S, Ganiats TG, Gelzer A, Hamilos D, Haydon RC 3rd, Hudgins PA, Jones S, Krouse HJ, Lee LH, Mahoney MC, Marple BF, Mitchell CJ, Nathan R, Shiffman RN, Smith TL, Witsell DL. Clinical practice guideline: adult sinusitis. Otolaryngol Head Neck Surg. 2007 Sep;137(3 Suppl):S1-31. doi: 10.1016/j.otohns.2007.06.726. PMID 17761281
- [Derived] Lehmann AE, Raquib AR, Siddiqi SH, Meier J, Durand ML, Gray ST, Holbrook EH. Prophylactic antibiotics after endoscopic sinus surgery for chronic rhinosinusitis: a randomized, double-blind, placebo-controlled noninferiority clinical trial. Int Forum Allergy Rhinol. 2021 Jul;11(7):1047-1055. doi: 10.1002/alr.22756. Epub 2020 Dec 19. PMID 33340285

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 134 participants signed consent, but only 89 were randomized. The remainder failed screening.
Period: Overall Study
Arm/Group | Amoxicillin-Potassium Clavulanate | Placebo
Started | 43 | 46
Completed | 38 | 41
Not Completed | 5 | 5
Not completed — Lost to Follow-up | 2 | 4
Not completed — Physician Decision | 1 | 0
Not completed — Protocol Violation | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Amoxicillin-Potassium Clavulanate | Placebo | Total
Number analyzed (Participants) | 38 | 41 | 79
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 37 | 40 | 77
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Full Range); unit: years] | 46.5 [18.5 to 67.3] | 40.8 [21.8 to 67.1] | 43.65 [18.5 to 67.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 27
  Male | 24 | 28 | 52
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 38 | 41 | 79
Lund Kennedy Endoscopic Score [Mean (Full Range); unit: units on a scale] — The Lund Kennedy endoscopic score is a grading system for visually evaluating patient's sinus cavities before and after surgery. It has five measures to score (polyps, edema, discharge, scaring, and crusting).
  Scores range from 0 to 20 with higher scores indicating greater sinus disease.
  units on a scale | 8.2 [4 to 14] | 8.2 [1 to 14] | 8.2 [1 to 14]
SNOT-22 Scores [Mean (Full Range); unit: units on a scale] — The sinonasal outcome test -22 (SNOT-22) is a validated instrument for measuring quality of life outcomes in chronic sinusitis.
  Snot-22 scores can range from 0 to 110. Higher scores indicate more severe symptoms.
  units on a scale | 47.8 [0 to 93] | 39.0 [10 to 84] | 43.4 [0 to 93]

OUTCOME MEASURES:

1. Primary Outcome: Sinonasal Outcome Test - 22
Description: The sinonasal outcome test -22 (SNOT-22) is a validated instrument for measuring quality of life outcomes in chronic sinusitis.
  Snot-22 scores can range from 0 to 110. Higher scores indicate more severe symptoms.
Time Frame: One week post operatively
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Amoxicillin-Potassium Clavulanate | Placebo
Number analyzed (Participants) | 38 | 41
score on a scale | 31.3 (21.7) | 31.0 (19.4)

2. Primary Outcome: Sinonasal Outcome Test - 22
Description: as for outcome 1
Time Frame: Six weeks post operatively
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Amoxicillin-Potassium Clavulanate | Placebo
Number analyzed (Participants) | 38 | 41
score on a scale | 22.3 (21.5) | 17.5 (15.3)

3. Secondary Outcome: Lund Kennedy Endoscopic Score
Description: The Lund Kennedy endoscopic score is a grading system for visually evaluating patient's sinus cavities before and after surgery. It has five measures to score (polyps, edema, discharge, scarring, and crusting).
  Scores range from 0 to 20 with higher scores indicating greater sinus disease.
Time Frame: One week postoperatively
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Amoxicillin-Potassium Clavulanate | Placebo
Number analyzed (Participants) | 38 | 41
score on a scale | 5.6 (1.8) | 5.9 (2.9)

4. Secondary Outcome: Lund Kennedy Endoscopic Score
Description: as for outcome 3
Time Frame: Six weeks postoperatively
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Amoxicillin-Potassium Clavulanate | Placebo
Number analyzed (Participants) | 38 | 41
score on a scale | 4.3 (2.6) | 4.5 (2.8)

5. Other Pre Specified Outcome: Number of Participants With Post Operative Infection
Description: The investigators will record the rate of post operative infections in the two groups.
Time Frame: One week postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Amoxicillin-Potassium Clavulanate | Placebo
Number analyzed (Participants) | 38 | 41
Participants | 1 | 0

6. Other Pre Specified Outcome: Number of Participants With Post Operative Infection
Description: The investigators will record the rate of post operative infections in the two groups.
Time Frame: Six weeks postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Amoxicillin-Potassium Clavulanate | Placebo
Number analyzed (Participants) | 38 | 41
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Follow-ups at one week post-surgery and then 6 weeks post-surgery
Arm/Group | Amoxicillin-Potassium Clavulanate | Placebo
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/46
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/46
Other Adverse Events (participants affected / at risk) | 10/43 | 1/46
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amoxicillin-Potassium Clavulanate (N=43) | Placebo (N=46)
Diarrhea (Gastrointestinal disorders) | 9 (9) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2014-10-06): https://cdn.clinicaltrials.gov/large-docs/11/NCT01919411/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-28): https://cdn.clinicaltrials.gov/large-docs/11/NCT01919411/SAP_002.pdf